CLINICAL TRIAL: NCT05005949
Title: STOP Persistent AF Post-Approval Study, a Sub-study to the Cryo Global Registry
Brief Title: STOP Persistent AF PAS
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: STOP Persistent AF PAS
Record Dates: First submitted 2021-07-29; First posted 2021-08-16 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Arctic Front™ Cardiac Cryoablation Catheter System — Pulmonary vein isolation will be performed with the Arctic Front™ Cardiac Cryoablation Catheter System

SUMMARY:
The STOP Persistent AF Post Approval Study (PAS) is a prospective, global, multicenter, observational trial.

DETAILED DESCRIPTION:
The STOP Persistent AF Post Approval Study (PAS) is a sub-study to the Cryo Global Registry. The PAS is a prospective, global, multicenter, observational trial. The purpose of the PAS is to describe long-term clinical performance and safety data in the Persistent AF population treated with Arctic Front™ and Freezor™ MAX Families of Cardiac Cryoablation Catheters (hereafter referred to as Arctic Front™ Cardiac Cryoablation Catheter System). This PAS is a condition of the Pre-Market Approval order (P100010/S098) by the U.S. Food and Drug Administration. Up to 400 subjects will be enrolled to ensure 355 are treated. A minimum of 50% of patients will be enrolled and treated in the US. The follow-up duration for this post-approval study will be 36-months.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with persistent AF.
* Subject is ≥ 18 years of age or minimum age as required by local regulations.
* Planned pulmonary vein isolation (PVI) procedure using commercially available Arctic Front™ Cardiac Cryoablation Catheter System.
* Willing to comply with study requirements and give informed consent (defined as legally effective, documented confirmation of a subject's voluntary agreement to participate in this clinical study) or authorization per institution and geographical requirements.

Exclusion Criteria:

* Subject has had a prior atrial ablation (except for cavo-tricuspid isthmus (CTI) ablation for AFL).
* Subject is enrolled in a concurrent study that has not been approved for concurrent enrollment by the global study manager.
* Subject with exclusion criteria required by local law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years of age (or minimum age as required by local regulations) who have a recommendation for a pulmonary vein ablation with the Arctic Front™ Cardiac Cryoablation Catheter System may be approached regarding enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial Fibrillation (AF) /Atrial Flutter (AFL) /Atrial Tachycardia (AT) | 36 months
  Estimate the 36-month freedom from Atrial Fibrillation (AF) /Atrial Flutter (AFL) /Atrial Tachycardia (AT) recurrence using the Arctic Front™ Cardiac Cryoablation Catheter System.
Freedom from Primary Safety Events | 12 months
  Estimate primary safety Adverse Event (AE) rates for cryoablation using the Arctic Front™ Cardiac Cryoablation Catheter System through 12-months.

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Tarakji, MD, Study Director — Medtronic CAS Chief Medical Officer
Locations (17):
- United States (10):
  - Hartford Hospital, Hartford, Connecticut
  - Cardiology Associates of Fairfield County, Stamford, Connecticut
  - BayCare Medical Group Cardiology, Clearwater, Florida
  - Heart Rhythms Solutions, Davie, Florida
  - Carle Foundation Hospital, Urbana, Illinois
  - Henry Ford Heart & Vascular, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - The Lindner Research Center, Cincinnati, Ohio
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Texas Health Research & Education Institute, Dallas, Texas
- Kepler Universitätsklinikum Med Campus III., Linz, Austria
- Germany (3):
  - St. Vinzenz-Hospital Köln, Cologne
  - MVZ CCB Frankfurt und Main Taunus, Frankfurt am Main
  - Städtische Kliniken München GmbH - Klinikum Bogenhausen, München
- Universitaria Pisana - Stabilimento di Cisanello, Pisa, Italy
- Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodz, Lodz, Poland
- Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool, United Kingdom